CLINICAL TRIAL: NCT00267033
Title: Randomized Trial of Vertebroplasty and Radiotherapy Versus Radiotherapy Alone for Osseous Spine Metastases
Brief Title: Evaluation of Vertebroplasty Associated With Radiotherapy for Spine Metastases (EVAR)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Myriem CARRIER, Department Clinical Research of Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P040426; AOM04013
Record Dates: First submitted 2005-12-19; First posted 2005-12-20 (Estimated); Last update posted 2008-12-02 (Estimated); Status verified 2007-03

CONDITIONS: Osseous Spine Metastases
Keywords: Neoplasm Metastasis; Bone Neoplasms; Pain; Radiotherapy; Vertebroplasty; Combined modality therapy
MeSH Terms: conditions — Neoplasm Metastasis; Bone Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): injection of orthopaedic cement into vertebral bodies
  Interventions: Procedure: injection of orthopaedic cement into vertebral bodies

INTERVENTIONS:
Procedure: injection of orthopaedic cement into vertebral bodies — injection of orthopaedic cement into vertebral bodies

SUMMARY:
A randomized phase III study of palliative external beam radiotherapy (RTOG 97-14) has shown that 8 Gy in a single fraction is very effective in providing pain relief, with complete or partial improvement in pain seen in 66% of patients with bone metastases. Percutaneous vertebroplasty (PV) is a technique designed to consolidate pathologic vertebral bodies through the injection of orthopaedic cement under fluoroscopic guidance. Consolidation provides rapid pain relief to painful vertebral body lesions secondary to osteoporosis, haemangiomas, myeloma and metastatic diseases, with complete or partial improvement in pain seen in 70-85% of patients. To date, no randomized trial has tested the association of vertebroplasty and radiotherapy to enhance pain relief for patients with painful osseous spine metastases.

A randomized trial has been designed to determine whether vertebroplasty and radiotherapy (8 Gy in a single fraction) provide enhancement pain and narcotic relief compared to radiotherapy alone for patients with painful osseous spine metastases

DETAILED DESCRIPTION:
Patients with 1 to 4 painful osseous spine metastases are randomized to 1 of 2 treatment arms:

* Arm 1: 8 Gy in a single fraction
* Arm 2: 8 Gy in a single fraction followed by vertebroplasty of the vertebral bodies, within 14 days after radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Osseous spine metastases from squamous cell carcinoma or adenocarcinoma
* One to four painful metastases located between the second cervical vertebra and the fifth lumbar vertebra
* Moderate to severe pain
* No spinal cord compression
* Karnofsky performance status > 40

Exclusion Criteria:

* Previous radiotherapy or surgery
* Vertebral fracture or any other formal indication of stabilization of the rachis by surgery or vertebroplasty
* Spinal cord compression
* Known anomaly of the haemostasis, or needed anticoagulant treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2005-11; Primary Completion 2008-02 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain relief with the Brief Pain Index (BPI), by a blind arm trial algologist, 3 months after radiotherapy. | 3 months after radiotherapy
Response will be scored as complete (no pain), partial (improvement of < 2 points in BPI), stable (+/- 1 point change in BPI) or progressive (> 2 point worsening of BPI). | during the study
Complete and partial responses will be considered treatment success, and stable and progressive responses will be considered treatment failures | during the study

SECONDARY OUTCOMES:
Evaluation of pain relief one month after radiotherapy | one month after radiotherapy
BPI-SF and EORTC QLQ-C30 will be used to assess general cancer quality of life. | during the study
The incidence of vertebral pathologic fracture will be registered. | one month after radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: jean-Marc SIMON, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- CHU Pitié-Salpétrière, Paris, France

REFERENCES:
- [Background] Hartsell WF, Scott CB, Bruner DW, Scarantino CW, Ivker RA, Roach M 3rd, Suh JH, Demas WF, Movsas B, Petersen IA, Konski AA, Cleeland CS, Janjan NA, DeSilvio M. Randomized trial of short- versus long-course radiotherapy for palliation of painful bone metastases. J Natl Cancer Inst. 2005 Jun 1;97(11):798-804. doi: 10.1093/jnci/dji139. PMID 15928300
- [Background] Weill A, Chiras J, Simon JM, Rose M, Sola-Martinez T, Enkaoua E. Spinal metastases: indications for and results of percutaneous injection of acrylic surgical cement. Radiology. 1996 Apr;199(1):241-7. doi: 10.1148/radiology.199.1.8633152.